CLINICAL TRIAL: NCT00942851
Title: A Study of Acetyl Hexapeptide-8 (AH8) in Treatment of Blepharospasm
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: BCN Peptides (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 090193; 09-N-0193
Record Dates: First submitted 2009-07-18; First posted 2009-07-21 (Estimated); Results first posted 2012-09-06 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-08

CONDITIONS: Focal Dystonia
Keywords: Dystonia; Blepharospasm; Botulinum Toxin; Treatment; Clinical Trial; Focal Dystonia
MeSH Terms: conditions — Dystonic Disorders; Dystonia; Blepharospasm

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- active (Experimental): AH-8 containing topical intervention
  Interventions: Drug: Acetyl-Hexapeptide Topical Treatment
- placebo (Placebo Comparator): topical intervention WITHOUT AH-8
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Acetyl-Hexapeptide Topical Treatment — AH-8 containing topical treatment
  Arms: active
Drug: placebo — topical treatment NOT containing AH-8
  Arms: placebo

SUMMARY:
Background:

* Blepharospasm is caused by excessive contraction of the muscles that close the eye. It can be treated with injections of botulinum neurotoxin (BoNT), which works by weakening those muscles.
* Acetyl Hexapeptide-8 (AH-8) is the active ingredient in a number of cosmetic creams used to treat wrinkles, and is marketed under the trade name Argireline(Copyright). Like BoNT, AH-8 works to weaken the muscles, but is available as a skin cream instead of an injection. AH-8 has never been used to treat people with blepharospasm.

Objectives:

- To determine if AH-8 can be used as part of a treatment regimen for blepharospasm.

Eligibility:

- Individuals 18 years of age and older who have blepharospasm and have been receiving successful treatment with botulinum toxin injections.

Design:

* Participants will be involved in the study for a maximum of 7 months.
* Patients will have a complete physical and neurological exam, and will be asked questions about their blepharospasm. Patients will then receive BoNT injections in the same areas of the muscle around the eye and at the same doses that have been effective previously.
* After the injections, patients will receive a container of either the active cream (with AH-8) or cream without AH-8, and will be instructed on how to apply it.
* Patients will return 1 month after the first visit for another neurologic exam and questions, and will be asked about any side effects. Another supply of cream will be given.
* Five additional visits will take place on a monthly basis, and patients will be given additional supplies of the cream as needed. Patients will stop participating in the study if they require another BoNT injection for blepharospasm. The study will end after 7 months.

DETAILED DESCRIPTION:
OBJECTIVE:

To study the efficacy of cutaneous application of Acetyl Hexapeptide-8 (AH8) in the therapy of blepharospasm.

STUDY POPULATION:

22 patients with blepharospasm.

DESIGN:

This will be a double blind, placebo-controlled trial. Patients receiving treatment of blepharospasm with botulinum neurotoxin (BoNT) will be recruited. They will receive either the study substance or a placebo cream containing the emulsion but no active substance, in twice daily applications to the eyelids beginning the day following a BoNT injection treatment. They will continue to apply the cream and we will record the time until their condition worsens back to baseline following benefit from the injections, hypothesizing that the cream application will prolong the time until the need for the next injection by at least 3 months.

OUTCOME MEASURES::

Primary: time until the Jankovic Blepharospasm Rating Scale (JBRS) reverts back to baseline.

Secondary: Change in the JBRS at 6 months; Change in the JBRS at 7 months if not receiving BoNT; Change in the JBRS at 3 months; Change in the Blepharospasm Disability Scale at 6 months

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age above 18 years
  2. Diagnosis of PB made by a Movement Disorders Neurologist
  3. Severity of PB prompting the need for treatment as determined by patient subjective assessment.
  4. JBRS of at least 3 at initial visit.
  5. BDS of at least 8 at the entry visit.
  6. At least three prior successful injectable BoNT treatments, with stable interval between injections of 3 months (ie duration of response of 3 months).

EXCLUSION CRITERIA:

1. Pregnant women
2. Blepharospasm associated with a different Neurologic condition, including but not limited to generalyzed dystonia, a parkinsonian syndrome, or major brain structural abnormality, as evidenced by Neurologic exam and/or review of records
3. Skin condition resulting in loss of integrity of the skin overlying the OO or potentially interfering with cream absorption.
4. Medical condition impairing the patient's ability to comply with the study protocol or to perform daily applications of the cream as instructed
5. Abnormally long or short response to BoNT treatment in the past, ie duration of PB relief with BoNT greater than 4 months or less than 2 months.
6. Allergy to any component of the study or placebo cream.
7. Known or observed eye pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ben Simon GJ, McCann JD. Benign essential blepharospasm. Int Ophthalmol Clin. 2005 Summer;45(3):49-75. doi: 10.1097/01.iio.0000167238.26526.a8. No abstract available. PMID 15970766
- [Background] Defazio G, Livrea P. Primary blepharospasm: diagnosis and management. Drugs. 2004;64(3):237-44. doi: 10.2165/00003495-200464030-00002. PMID 14871168
- [Background] Defazio G, Livrea P. Epidemiology of primary blepharospasm. Mov Disord. 2002 Jan;17(1):7-12. doi: 10.1002/mds.1275. PMID 11835433

RESULTS

PARTICIPANT FLOW:
Groups:
- Active: Topical intervention agent containing AH8 0.005% Twice daily application to the eyelids in standardized fashion.
- Placebo: Topical intervention agent WITHOUT AH-8. Identically appearing cream without the active ingredient.
  Twice daily application to the eyelids in standardized fashion.
Period: Overall Study
Arm/Group | Active | Placebo
Started | 12 | 12
Completed | 12 | 11
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 2 | 1 | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 57.59 (8.46) | 55.87 (8.25) | 56.73 (8.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 2 | 14
  Male | 0 | 10 | 10
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Time Until Jankovic Blepharospasm Rating Scale (JBRS) Reverts Back to Baseline
Description: The JBRS is a severity scale for blepharospasm, ranging from 0 (no symptoms) to 8 (the most severe symptoms, functionally blind). It includes measures of blink frequency and severity of abnormal eye closure. The scale was measured at baseline (before intervention) and followed over time. Return to baseline value represents loss of benefit from BoNT injection. The time to return to baseline JBRS is an indication of added benefit from the topical intervention.
Time Frame: 3-7 months
Measure: Mean (Standard Deviation); unit: month
Groups:
- Active Ingredient- AH8: subjects receiving active intervention, ie topical cream containing 0.005% AH-8
- Placebo: subjects receiving placebo intervention, ie identically-appearing topical cream without AH-8 content
Arm/Group | Active Ingredient- AH8 | Placebo
Number analyzed (Participants) | 12 | 11
month | 3.71 (1.48) | 3.03 (.23)

2. Secondary Outcome: Change in the JBRS at 3 Months
Description: The JBRS is a severity scale for blepharospasm, ranging from 0 (no symptoms) to 8 (the most severe symptoms, functionally blind). It includes measures of blink frequency and severity of abnormal eye closure. The scale was measured at baseline (before intervention) and followed over time.
Time Frame: baseline to 3 months
Population: One placebo arm participant dropped out due to unrelated personal problems
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Active Ingredient- AH8 | Placebo
Number analyzed (Participants) | 12 | 11
points | 1.09 (0.7) | 0.92 (2.07)

3. Secondary Outcome: % Blepharospasm Disability Scale (BDS) Change at 3 Months
Description: % BDS change at 3 months. The BDS is a quality of life scale ranging from 0 (no symptoms) to 26 (maximum impact of symptoms on quality of life). The questions are specific for impairment related to blepharospasm. We compared the percentage change over three months in the active and placebo arms.
Time Frame: baseline to 3 months
Population: One placebo arm participant discontinued study due to unrelated personal problems
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Active | Placebo
Number analyzed (Participants) | 12 | 11
percentage change | 30.89 (37.3) | 32.32 (31.13)

ADVERSE EVENTS:
Arm/Group | Active | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=12) | Placebo (N=12)
eyelid irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) — 4 subjects (2 active arm and 2 placebo arm) experience minor self-limited eyelid irritation. Ophthalmology consultation was obtained in all cases. No change in the study procedure was needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes